CLINICAL TRIAL: NCT02067169
Title: A French Cohort of Transplant Recipients With CMV Infection : Risk Factors for Antiviral Resistance in the Prophylaxis Era. Survey of Pharmacological and Virological Resistance of Cytomegalovirus to Antiviral Therapy in Transplantation.
Brief Title: A French Cohort of Transplant Recipients With CMV Infection : Risk Factors for Antiviral Resistance in the Prophylaxis Era.
Acronym: ORPHAVIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09013 ORPHAVIC
Record Dates: First submitted 2014-02-14; First posted 2014-02-20 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Transplant Recipients With CMV Infection
Keywords: Transplantation; CMV infection; antiviral resistance
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Detection of the CMV in sang, the leukocytes, or plasma with or without the viral quantification and/or the sample of urine of saliva or tissues, positive for research of CMV.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CMV infection: allograft recipient with active CMV infection
  Interventions: Biological: CMV Infection

INTERVENTIONS:
Biological: CMV Infection — Routine follow-up (viral load, creatininaemia, neutrophil count, isolation of CMV strains when possible) and biological sample collection for . Resistance testing towards any antiviral available by genotype and phenotype (when an isolate is obtained) when resistance criteria are fulfilled. Plasma collection at treatment initiation, and in case of neutropenia, for antiviral dosage.

SUMMARY:
Resistance to antivirals is a growing problem in transplantation.that may concerns up to 5% of patients treated for cytomegalovirus (CMV) syndrome or disease in recent per-protocol studies. This prevalence vary with the organ transplanted and the degree of viral replication and immunosuppression. Less data are available to date from real-life cohorts of patients, and there is no systematic survey of resistance in Europe or in the US. Non response to treatment concerns a larger group of patients and can result either from emergence of a resistant strain (virological resistance), from inadequate dosage of antivirals, or a high degree of immunosuppression, with a poor CMV immune response. The respective clinical impact of virological resistance and clinical resistance (of pharmacological or immunological origin) on graft outcome and long-term survival of patients has never been assessed. High viral loads and persistent replication associated to prolonged exposure to antivirals are known to favor the emergence of resistant strains. Though epidemiology of resistant strains, role of multiple infections, impact of various mutations on degree of resistance to antivirals and outcome remains to be further studied. Most studies are per-protocol studies or short-term studies conducted on limited populations. There are no data in real-life of transplanted patients at the era of enlarged prophylaxis except those from the French survey for cytomegalovirus resistance cohort opened at the end of 2006. From the first data collected on 346 patients we shown a 10,6% prevalence of non-response to therapy with 5,2% of virological resistance (6,1% incidence at one year on 214 patients) with a trend to poorer outcome in case of virological resistance and to the absence of impact of prophylaxis versus preemptive therapy, though larger populations and prolonged follow-up are requested to fulfill all objectives.

We therefore aim to constitute a prolonged survey cohort for CMV resistance with a large number of patients and a prolonged follow-up, to gather data on resistance to antivirals in real-life of transplant patients in an organized data bank, This cohort is in the continuum of our previous cohort started in 2006, granted by the Hospital Clinical Research Program Interregional (PHRC), with the same major objectives and prolonged follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* allograft recipient with active CMV infection,
* or patient from the previous cohort, without opposition to biological collection of samples

Exclusion Criteria:

* not willing to participate, no health insurance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: allograft recipient or hematopoietic stem cell or solid organ.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
prevalence and incidence of resistance of cytomegalovirus | 3 weeks
  Non response to therapy is defined as persistent viral replication after more than 3 weeks of appropriate antiviral treatment, with or without clinical manifestations.

SECONDARY OUTCOMES:
pharmacological and virological resistance | 2 years
  Measure the respective incidence of pharmacological and virological resistance

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ALAIN, MD, Principal Investigator — Limoges UH
Locations (38):
- France (38):
  - Virologie, Amiens
  - Virologie, Angers
  - Virologie, Besançon
  - Virologie - Hôpital Avicenne, Bobigny
  - Virologie, Bordeaux
  - Virologie, Brest
  - Virologie, Caen
  - Virologie, Clermont-Ferrand
  - AP-HP - Hôpital Beaujon - Virologie, Clichy
  - AP-HP - Hôpital MONDOR - Virologie, Créteil
  - Virologie, Dijon
  - Virologie, Grenoble
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Virologie, Lille
  - Bactériologie Virologie, Limoges
  - HCLYON - Virologie - Hôpital La Croix Rousse, Lyon
  - Virologie, Lyon
  - Virologie - AP-HM - La Timone, Marseille
  - Virologie, Montpellier
  - Virologie, Nancy
  - Virologie, Nantes
  - Virologie, Nîmes
  - AP-HP - Hôpital Saint-Antoine - Virologie, Paris
  - AP-HP - Hôpital Georges Pompidou - Virologie, Paris
  - AP-HP - Hôpital TENON - Virologie, Paris
  - Virologie - Hôpital BICHAT, Paris
  - Virologie - Hôpital La Pitié Salpétrière, Paris
  - Virologie - Hôpital NECKER, Paris
  - Virologie - Hôpital SAINT-LOUIS, Paris
  - Virologie, Poitiers
  - Virologie, Reims
  - Virologie, Rennes
  - Virologie, Rouen
  - Virologie, Saint-Etienne
  - Virologie, Strasbourg
  - Virologie, Toulouse
  - Virologie, Tours
  - Virologie - Hôpital Paul Brousse, Villejuif